CLINICAL TRIAL: NCT03975751
Title: A Survey on the Practice of Sedation and Analgesia Among Patients With Severe Brain Injury in China: a Prospective Observational Study
Brief Title: Practice of Sedation and Analgesia in Patients With Severe Brain Injury in China
Status: Completed | Type: Observational
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Jian-Xin Zhou, Professor, Capital Medical University
Other Study IDs: KY2017-062-02
Record Dates: First submitted 2019-06-02; First posted 2019-06-05 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Intensive Care Unit
Keywords: severe brain injuries; sedation and analgesia; intensive care unit; survey
MeSH Terms: conditions — Brain Injuries; Agnosia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: The Glasgow Coma Scale (GCS) — Use the common GCS, RASS and self-reported pain assessment for evaluating consciousness, agitation/sedation and analgesia.
  Other Names: The Richmond Agitation-Sedation Scale (RASS); The self-reported pain assessment

SUMMARY:
Sedation and analgesia is necessary management for patients in the intensive care units. The high-level studies of sedation and analgesia in China are still deficient, especially in patients with brain injuries who even have been excluded from the relevant studies.

DETAILED DESCRIPTION:
Sedation and analgesia is necessary management for patients in the intensive care units. The high-level studies of sedation and analgesia in China are still deficient, especially in patients with brain injuries who even have been excluded from the relevant studies. In the present study, a multicenter, 1-day point cross-sectional study about the sedation and analgesia among patients in China, particularly brain-injured will be investigated. The objectives are to investigate sedation and analgesia among patients in China and to compare sedation and analgesia between brain injuries and other patients.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients admitted to the participating ICUs on the investigation day

Exclusion Criteria:

* Age under 18 years
* Less than 24 hours of ICU stay before screening
* Taking part in other studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the patients at 9am on the on-site investigation day in the participating ICUs will be screened and enrolled according to the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 387 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2019-01-08 (Actual); Study Completion 2019-03-09 (Actual)

PRIMARY OUTCOMES:
Performance of sedation assessment | The previous 24 hours prior to the on-site investigation
  The percentage of patients receiving sedation assessment
Performance of pain assessment | The previous 24 hours prior to the on-site investigation
  The percentage of patients receiving pain assessment

SECONDARY OUTCOMES:
Use of sedatives | The previous 24 hours prior to the on-site investigation
  The percentage of patients receiving sedatives
Use of analgesics | The previous 24 hours prior to the on-site investigation
  The percentage of patients receiving analgesics
ICU mortality | Within 60 days after on-site investigation
  The percentage of patients dead in the ICU
Hospital mortality | Within 60 days after on-site investigation
  The percentage of patients dead in the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Jian-Xin Zhou, MD, Study Chair — Beijing Tiantan Hospital
Locations (1):
- ICU, Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chen K, Yang YL, Li HL, Xiao D, Wang Y, Zhang L, Zhou JX. A gap existed between physicians' perceptions and performance of pain, agitation-sedation and delirium assessments in Chinese intensive care units. BMC Anesthesiol. 2021 Feb 25;21(1):61. doi: 10.1186/s12871-021-01286-w. PMID 33627067